CLINICAL TRIAL: NCT01968811
Title: A Multi-Centre, Post CE Mark, Open Clinical Investigation to Evaluate an Abdominal NPWT (Negative Pressure Wound Therapy) System (Avance® Pump and Avance® Foam Abdominal Dressing Kit) in Subjects With Open Abdominal Wounds
Brief Title: Post Market Clinical Follow Up Study of Avance Foam Abdominal Dressing Kit in Open Abdomen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Avance A01
Record Dates: First submitted 2013-10-14; First posted 2013-10-24 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2014-05

CONDITIONS: Open Abdomen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avance foam, abdominal dressing kit (Experimental)
  Interventions: Device: Avance Foam dressing kit

INTERVENTIONS:
Device: Avance Foam dressing kit

SUMMARY:
The investigation is a Post Marketing Follow-Up Study for the Avance Foam Abdominal Dressing Kit conducted as part of Mölnlycke Health Care's quality system. The primary objective is to evaluate the dressing kit as part of a negative pressure system. The secondary objectives are to collect and evaluate safety data, performance data and information on technical complications.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent from subject or family member
2. Subjects with open abdomen suitable for temporary closure with NPWT therapy
3. Subjects where the viscera and/or abdominal organs need to be protected by an abdominal organ contact layer (OCL)
4. Subject which (at the time of the baseline visit) are planned to be cared for between dressing changes at Intensive Care Unit
5. Male or female, 18 years and above

Exclusion Criteria:

1. Synthetic mesh inserted in the abdomen
2. Non-enteric fistulae or unexplored fistulas
3. Untreated osteomyelitis
4. Malignant wounds
5. Abdominal wall hernia
6. Subjects previously treated with an NPWT abdominal dressing
7. Known allergy or hypersensitivity to any of the components in the dressing
8. Pregnancy
9. Subjects not suitable for the investigation according to the investigator's judgement
10. Subjects included in other ongoing clinical investigation at present which could interfere with this investigation, as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University hospital, Gothenburg, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Avance Foam, Abdominal Dressing Kit: Avance Foam dressing kit
Period: Overall Study
Arm/Group | Avance Foam, Abdominal Dressing Kit
Started | 10
Completed | 5
Not Completed | 5
Not completed — Protocol Violation | 4
Not completed — post op.ref. of subject to other hospita | 1

BASELINE CHARACTERISTICS:
Arm/Group | Avance Foam, Abdominal Dressing Kit
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  Sweden | 10

OUTCOME MEASURES:

1. Secondary Outcome: - Fascial/Skin Closure of the Open Abdomen
Description: The performance objective is assessed through general application and removal questions after each investigational device handling.
Time Frame: End of treatment, up to 4 days.
Population: No. Analysed for efficacy ITT 10 , PP 9,
Measure: Number; unit: participants
Arm/Group | Avance Foam, Abdominal Dressing Kit
Number analyzed (Participants) | 10
participants
  Closed fascia | 5
  insertion of synthetic mesh | 3

2. Primary Outcome: To Evaluate the Performance of the Dressing Kit as Part of a Negative Pressure System in Post Market Clinical Follow-up Settings
Description: Outcome of each subject was evaluated and presented individually. Questionnaires answered by surgeon at application and removal of the kit; Baseline Overall ease of application of the kit: No. of surgeons rated as; Very easy= 4/Easy=3/Somewhat easy=2/Not easy Overall satisfaction with the kit:No. of surgeons rated as Very satisfied=3/ Satisfied=5/ Unsatisfied=2/ Very unsatisfied=0
  Questionnaires were answered by surgeon at application and removal of the kit; Visit 2 Overall ease of application of the kit:No.of surgeons rated as Very easy= 2/Easy=5/Somewhat easy=0/Not easy=1 Overall satisfaction with the kit: No.of surgeons rated as Very satisfied=1/ Satisfied=3/ Unsatisfied=4/ Very unsatisfied=0 Visit 3 Overall ease of application of the kit: No.of surgeons rated as Very easy= 0/Easy=6/Somewhat easy=0/Not easy=0 Overall satisfaction. No of surgeons rated as Very satisfied=0, satisfied=4, unsatisfied=2, very unsatisfied=0
Time Frame: From 1 to 3 visit, depending on each subject/wound, up to 4 days.
Population: 10 patients were enrolled and individually analysed and presented in the study
Measure: Number; unit: number of surgeons
Arm/Group | Avance Foam, Abdominal Dressing Kit
Number analyzed (Participants) | 10
number of surgeons
  ease of application Very easy | 4
  Ease of application Easy | 3
  Ease of application Some what easy | 2
  Ease of application Not easy | 1
  Overall satisfaction with the kit, Very satisfied | 3
  Overall satisfaction with the kit, Satisfied | 5
  Overall satisfaction with the kit, Unsatisfied | 2

ADVERSE EVENTS:
Arm/Group | Avance Foam, Abdominal Dressing Kit
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avance Foam, Abdominal Dressing Kit (N=10)
OCL migration (General disorders) | 3 (3)
bowel ischemia (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avance Foam, Abdominal Dressing Kit (N=10)
blistering of skin (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No